CLINICAL TRIAL: NCT05320354
Title: Diagnosis and Bacterial Identification of Periprosthetic Joint Infection With Microbial-ID
Acronym: MID
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: UMC Utrecht (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Principal Investigator, Harrie Weinans, Prof. Dr., UMC Utrecht
Other Study IDs: 22-072
Record Dates: First submitted 2022-04-01; First posted 2022-04-11 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Periprosthetic Joint Infection; PJI
Keywords: Microbial-ID test; Periprosthetic joint infection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients suspected of PJI: Adult patients, both male and female, scheduled for a puncture or surgery of their prosthetic joint due to suspected PJI.
  Interventions: Diagnostic Test: Microbial ID test

INTERVENTIONS:
Diagnostic Test: Microbial ID test — In addition to the standard of care procedure for patients suspected for a periprosthetic joint infection, the MID-test will be performed using the residual synovial fluid. Individual test results of the MID-test are not reported back to the participating sites in order to not interfere with the sites' standard of care approach.
  Other Names: Synovasure® Microbial Identification Test; Synovasure® Microbial ID P. acnes Test.

SUMMARY:
The primary objective of this study is to demonstrate the validity of the Microbial- ID test to aid in diagnosis of periprosthetic joint infection (PJI) in terms of sensitivity and specificity.

DETAILED DESCRIPTION:
In the diagnosis of periprosthetic joint infection (PJI) there is no golden standard test. Multiple definitions for the diagnosis of PJI exist, such as the European Bone and Joint Infection Society (EBJIS)1, Musculoskeletal Infection Society (MSIS)2, and the Infectious Diseases Society of America (IDSA)3. One of the criteria that defines PJI is that there are at least two positive periprosthetic cultures with phenotypically identical organisms. Although these two positive bacterial cultures can certainly be considered proof of PJI, many other criteria are also used, such as a sinus tract, white blood count (WBC), elevated C-reactive protein and/or erythrocyte sedimentation rate (ESR), elevated percentage of neutrophils, and positive alpha defensin. Even when all these criteria are negative, a PJI cannot be excluded. Zimmer Biomet developed the Synovasure® Microbial-ID test that enables early and faster identification of microbial species through detection of microbial antigens responsible for infection.

This is an international multicenter, non-randomized, prospective, non-intervention clinical investigation.The primary objective of this study is to demonstrate the validity of the Microbial-ID test to aid in diagnosis of PJI in terms of sensitivity and specificity. The study population is adult patients with a potentially infected joint implant, who will undergo an articular puncture and/or surgery with harvesting of synovial fluid. In addition to the standard of care procedure for patients with a suspected PJI, the MID-test will be performed using the residual synovial fluid. Individual test results of the MID-test are not reported back to the participating sites in order to not interfere with the sites' standard of care approach.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Patients do not benefit from participating in this study. A separate diagnostic tool will run in parallel but this procedure will not interfere with the patient's current path of diagnostic work up nor will it have an effect on their treatment plan. The results will help the investigators to get more insight in the reliability of the MID-test to detect microbial antigens responsible for the PJI. There are no known disadvantages for the patients taking part in this research.

ELIGIBILITY:
Inclusion Criteria:

* Patient has complaints (pain, stiffness) about the prosthetic joint And has clinical features for joint infection at physical examination (swelling, redness, warm, sinus tract) AND has an elevated serum CRP (>10 mg/L)
* Patient is scheduled for a puncture AND/OR surgery, with harvesting of synovial fluid
* Patient ≥ 18 years of age
* Patient is competent, able, and willing to provide written informed consent

Exclusion Criteria:

* Treatment with antibiotics ≤2 weeks prior to puncture and/or surgery;
* Other obvious reason(s) for implant dysfunction, such as: fracture, an implant breakage, a malposition, and/or a tumour.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a potentially infected joint implant, who will undergo an articular puncture and/or surgery with harvesting of synovial fluid.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the MID-test | after 3 weeks
  Sensitivity of the MID-test based upon the number of subjects with a positive MID-test AND ≥1 positive microbiology culture(s) for the same bacterial species (true positives) and the number of subjects with a negative MID-test AND ≥1 positive microbiology culture(s) for one of the four bacterial species the MID-test is testing for (false negatives).
Specificity of the MID-test | after 3 weeks
  Specificity of the MID-test based upon the number of subjects with a negative MIDtest AND only negative microbiology cultures (true negatives) and the number subjects with a positive MID-test AND only negative microbiology cultures (false positives).

SECONDARY OUTCOMES:
Comparison of MID-test and the MB culture(s) regarding the time-to-result. | after 3 weeks
  Comparison of the time-to-result (elapsing hours between harvesting and test result) of the MID-test and the microbiology culture(s).
Rate of identification of bacterial species by the MID-test and the corresponding MB culture(s). | after 3 weeks
  Rate of identification of bacterial species by the MID-test and the corresponding microbiology culture(s).
Proportion of agreement between the MID-test and the diagnosis of PJI according to the EBJIS definition. | after 3 weeks
  Proportion of agreement between the MID-test and the diagnosis of PJI according to the EBJIS definition as assessed by a blinded investigator.
Rate of "false positives" in the reported low-grade PJIs at ≥1-year follow-up. | after 1 year
  Rate of "false positives" (MID test (+) and MB culture (-) at F0) in the reported low-grade (MB (-) and clinical signs (+)) PJIs at ≥1-year follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Harrie Weinans, Prof, MD, Principal Investigator — H.H.Weinans@umcutrecht.nl
Locations (6):
- Charité Universitätsmedizin Berlin, Berlin, Germany
- UMC Utrecht, Utrecht, Netherlands
- Hospitalar do Porto,, Porto, Portugal
- Valdoltra Orthopeadic Hospital,, Valdoltra, Slovenia
- Hospital Clinic Barcelona, Barcelona, Spain
- Universitätsspital Basel,, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided